CLINICAL TRIAL: NCT05940532
Title: A Single-arm Phase 2 Study of Sugemalimab and Chemotherapy as Induction Therapy in Unresectable and Stage III Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Trial of Sugemalimab and Chemotherapy in Unresectable Stage III NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HTOSG Lung 001
Record Dates: First submitted 2023-06-26; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: immunotherapy; chemotherapy; radiotherapy; surgery; non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sugemalimab; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional arm (Experimental): Patients will receive 3 cycles of induction therapy with sugemalimab and chemotherapy before curative local therapy.
  Interventions: Drug: Sugemalimab and Chemotherapy

INTERVENTIONS:
Drug: Sugemalimab and Chemotherapy — Chemotherapy: Paclitaxel 175mg/m2 D1, Carboplatin AUC=5 or DDP 75mg/m2 D1 for NSCLC; Pemetrexed 500mg/m2 D1, Carboplatin AUC=5 or DDP 75mg/m2 D1 for non-squamous NSCLC; intravenous infusion every 3 weeks, for up to four cycles.
  Sugemalimab: 1200 mg by intravenous infusion every 3 weeks, for up to 2 years.

SUMMARY:
The goal of this phase II, open-label, single-arm study is to evaluate the efficacy and safety of induction immunotherapy and chemotherapy followed by the multidisciplinary team (MDT)-guided radiotherapy or surgery in unresectable, stage III non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1.18 to 75 years old, both male and female;

2.ECOG score: 0-1;

3.Histopathologically or cytologically confirmed, stage III (AJCC 8th) non-small cell lung cancer;

4.Multidisciplinary team (MDT) discussion confirmed unresectable disease but can be treated by curative radiotherapy;

5.Measurable lesions available;

6.Major organ function is basically normal;

7.Estimated survival time is at least 6 months;

8.Non-surgically sterile female subjects of childbearing age must have a negative serum HCG test before inclusion.

Exclusion Criteria:

1. Histologically or cytologically confirmed mixed SCLC and NSCLC;
2. Subjects with driver gene mutations(EGFR mutation, ALK fusion, etc.);
3. Previous systemic anti-tumor therapy including immune checkpoint inhibitors for NSCLC;
4. Previous thoracic radiotherapy;
5. Subjects who participated in other clinical trials within 4 weeks or 5 drug half-lives(whichever is shorter) before the first dose;
6. Systemic immunostimulant therapy before the first dose;
7. Systemic immunosuppressive therapy before the first dose or were expected to require systemic immunosuppressive drugs during the study treatment;
8. Subjects with autoimmune diseases;
9. Other malignant tumors other than non-small cell lung cancer within 5 years before screening;
10. Known or suspected interstitial pneumonia;
11. Other moderate to severe lung diseases that may interfere with the detection or treatment of drug-related pulmonary toxicity and seriously affect respiratory function;
12. Severe cardiovascular and cerebrovascular diseases;
13. Clinically significant bleeding symptoms or significant bleeding tendency within 1 month before the first dose;
14. Arteriovenous thrombotic events within 3 months before the first dose;
15. Positive HIV test;
16. Active hepatitis B or C;
17. Evidence of active tuberculosis infection within 1 year before the first dose;
18. Serious infection within 4 weeks before the first dose;
19. History of attenuated live vaccination 28 days before the first dose or expected to receive attenuated live vaccination during the study;
20. Major surgeries other than diagnosis or biopsy within 28 days prior to the first dose;
21. Previous or planned allogeneic bone marrow transplantation or solid organ transplantation;
22. History of severe allergic reactions to other monoclonal antibodies/fusion proteins;
23. Allergic to any component of the randomized treatment regimen;
24. Female subjects who are pregnant, lactating, or planning to get pregnant during the study period;
25. Subjects who have a known history of psychotropic drug abuse, alcoholism, or drug abuse;
26. Presence of other conditions that, in the opinion of the investigator, would make participation in this clinical trial inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
ORR | From the initiation of the first dose to 3 years
  Objective response rate

SECONDARY OUTCOMES:
PFS | From the initiation of the first dose to 3 years
  Progression-free survival
OS | From the initiation of the first dose to 3 years
  Overall survival
iORR | From the initiation of the first dose to 3 years
  Objective response rate after induction therapy
AEs | From the initiation of the first dose to 90 days after the last dose
  Adverse events
Measurement of Quality of Life with EORTC QLQ-C30 questionnaire | From the initiation of the first dose to 3 years
  EORTC QLQ-C30 questionnaire minimum value: not at all (1); maximum: very much (4); higher scores means a worse outcome
Measurement of Quality of Life with EORTC QLQ-LC13 questionnaire | From the initiation of the first dose to 3 years
  EORTC QLQ-LC13 questionnaire minimum value: not at all (1); maximum: very much (4); higher scores means a worse outcome
Measurement of Quality of Life with EORTC EQ-5D-5L VAS questionnaire | From the initiation of the first dose to 3 years
  The EQ-5D-5L VAS records the respondent's self-rated health on a 10 centimeter (cm) vertical, visual analogue scale. It is rated by the respondent on a scale 0 to 100, with 0 being "the worst health you can imagine" and 100 being "the best health you can imagine"

CONTACTS AND LOCATIONS:
Overall Officials: Hui Wang, MD, Principal Investigator — the Department of Radiation Oncology; Huai Liu, MD, Principal Investigator — the Department of Radiation Oncology
Locations (1):
- Hunan Cancer Hospital, Changsha, China